CLINICAL TRIAL: NCT06810063
Title: Feasibility and Reliability of the Melbourne Assessment-2 (MA-2) for Telehealth
Status: Active, not recruiting | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Jill Heathcock, Professor, Division of Physical Therapy, Ohio State University
Other Study IDs: 2023B0100
Record Dates: First submitted 2025-01-24; First posted 2025-02-05 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-01

CONDITIONS: Cerebral Palsy; Hemiplegic Cerebral Palsy
Keywords: Assessment; Telehealth
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- In-person vs. telehealth assessment: Participants will be randomly assigned to in-person visit first or telehealth visit first. Both groups will complete both visits. Each visit requires about 20 minutes.
  Interventions: Other: Assessment only, no intervention

INTERVENTIONS:
Other: Assessment only, no intervention — Participants in this study complete two visits to test the agreement of telehealth and in person assessments of arm and hand movement.

SUMMARY:
The goals of this study:

1. Determine if a play based test of arm and hand movements is valid and reliable when conducted through telehealth for children with hemiplegic cerebral palsy.
2. Measure differences in parent, provider and child engagement when an assessment is conducted in-person compared to via telehealth.
3. Rate caregivers' overall impressions of procedures when an assessment is conducted in-person compared to telehealth.

Participants will attend two visits, one in person and one through telehealth. During each visit, the child will play with common toys. The sessions will be video recorded and scored using two standardized assessments, the Melbourne Assessment-2 (MA-2) and the Assisting Hand Assessment.

DETAILED DESCRIPTION:
After a child has a stroke, noticeable and lifelong developmental concerns emerge. One side of the body is typically much weaker, often impacting the arm/hand more than the leg/foot, so we focus on the arm/hand. The weakness is like adults with stroke, but in children, stroke impairs play, reaching for/holding toys, communication gestures, and whole-body movement. Because of this, most children with pediatric stroke will receive physical and/or occupational therapy throughout childhood. Traditionally, rehabilitation occurs with the child, caregiver and therapist meeting in person at clinics, homes, or schools. However, telehealth rehabilitation, where the therapist and patient meet virtually through a computer or tablet, has emerged a sustainable and accessible alternative. Telehealth also has the potential to improve access to quality treatments, improve health outcomes and reduce healthcare costs. One problem with telehealth rehabilitation is that few assessments have been validated for use in telehealth. In adults with stroke, researchers have identified several assessments for that work well via telehealth. Similarly, in children with one specific brain disease, researchers found that the results of one commonly used gross motor test are similar when delivered via telehealth compared to in-person. Unfortunately, there is no studied arm/hand assessment for children with stroke. This makes it hard to measure if telehealth rehabilitation changes arm/hand function. This proposal will test two playful arm/hand assessments via telehealth. Investigators will test 35 children (2-10 years old) twice (once in-person and once via telehealth) with the same assessment and compare the results. Investigators will use two well-established assessments, the Melbourne Assessment-2 and the Assisting Hand Assessment. Both assessments will be recorded- via camera (in-person) and secure videoconferencing (telehealth). Those recordings will then be scored by a therapist trained in the Melbourne Assessment and Assisting Hand Assessment. Investigators will compare the results of both assessments to see if the scores match.

ELIGIBILITY:
Inclusion Criteria:

* ages 2-10 years old
* hemiplegic cerebral palsy
* able to attend an in-person visit in the research lab OR live within 60 miles of the research lab
* able to attend a telehealth session with personal device

Exclusion Criteria:

* child or caregiver does not speak English
* unable to attend one in person visit and one telehealth visit within 1 month

Ages: 2 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children, ages 2-10 years old with hemiplegic Cerebral palsy
Sampling Method: Non-Probability Sample
Enrollment: 35 (Estimated)
Dates: Start 2023-09-29 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Melbourne Assessment-2 | 1 month
  Upper Extremity assessment, range 0-100, higher score indicates better outcomes.
Assisting Hand Assessment | 1 month
  Upper extremity assessment, range 0-100, higher score indicates better outcomes.

SECONDARY OUTCOMES:
Acceptability Intervention Measure | immediately after telehealth visit
  Evaluate acceptability of telehealth assessment, 4 questions rated on 5-point Likert scale from 1 (strongly disagree) to 5 (strongly agree). Reported as proportion of items rated at or above 4/5
Intervention Appropriateness Measure | immediately after telehealth visit
  Evaluate appropriateness of telehealth assessment, 4 questions rated on 5-point Likert scale from 1 (strongly disagree) to 5 (strongly agree). Reported as proportion of items rated at or above 4/5
Feasibility of Intervention Measure | immediately after telehealth visit
  Evaluate feasibility of telehealth assessment, 4 questions rated on 5-point Likert scale from 1 (strongly disagree) to 5 (strongly agree). Reported as proportion of items rated at or above 4/5

CONTACTS AND LOCATIONS:
Overall Officials: Jill Heathcock, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Wexner Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: Undecided